CLINICAL TRIAL: NCT04763343
Title: Ketamine Treatment of Youth Suicide Attempters for Fast Reduction of Severe Suicide Risk and Facilitation of Long-term Collaborative Clinical Engagement: A Double Blind Randomized Placebo Controlled Trial
Brief Title: Ketamine Treatment of Youth Suicide Attempters
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tatiana Falcone, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Tatiana Falcone, MD, Staff, Cleveland Clinic, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-154; 1R01MH125214-01 (NIH)
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind, Placebo Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Treatment + CAMS Therapy (Experimental)
  Interventions: Drug: Ketamine Hydrochloride; Behavioral: CAMS Therapy
- Saline Placebo Treatment + CAMS Therapy (Placebo Comparator)
  Interventions: Drug: Saline; Behavioral: CAMS Therapy

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine hydrochloride will be given as an intravenous infusion using a standard regimen given in most studies conducted: 0.5 mg/kg over 40 minutes. Ketamine infusions will be given every other day until either the subject reports clinician rated Scale for Suicidal Ideation (SSI) score of<4, and >50% decrease from baseline, and clinical assessment of patient not being suicidal for three consecutive pre-infusion ratings, or a maximum of six infusions have been given over the course of 2 weeks, or they have been discharged from the inpatient unit.
  Arms: Ketamine Treatment + CAMS Therapy
Drug: Saline — Subjects randomized to placebo will be administered a saline (0.9% sodium chloride) drip for 40 minutes. Saline placebo infusions will be given every other day until either the subject reports clinician rated Scale for Suicidal Ideation (SSI) score of<4, and >50% decrease from baseline, and clinical assessment of patient not being suicidal for three consecutive pre-infusion ratings, or a maximum of six infusions have been given over the course of 2 weeks, or they have been discharged from the inpatient unit.
  Arms: Saline Placebo Treatment + CAMS Therapy
Behavioral: CAMS Therapy — CAMS weekly sessions will also be started immediately as an inpatient at the start of the study while receiving ketamine or saline. CAMS will be continued weekly after the patient is discharged and followed up as an outpatient. Weekly CAMS sessions will be terminated after the subject, as an outpatient, has three consecutive outpatient CAMS sessions with an overall risk < 2 (# 6 on the SSF Core Assessment) along with a positive response regarding their thoughts/feelings and clinician indicating behavioral stability (suicidal behavior).

SUMMARY:
Ketamine, an NMDA antagonist, has been shown to have rapid anti- suicidal effects. However, its safety and efficacy and special populations has not been investigated and documented. Several reports in adults suggest rapid decrease of suicidal ideation. In the last decade there is an alarming increase of the number of suicide attempts in patients ages 14-30. Suicide is the second leading cause of death in this population. Patients with previous history of suicide attempt, are even in a higher risk category. The present study focus in this high risk group of suicide attempters. This will be a randomized controlled trial enrolling 60 youth between the ages 14-30 after a suicide attempt; patients will be randomized to receive Ketamine 0.5 mg/kg over 40 minutes or normal saline. Patients will receive all Ketamine or placebo infusions while admitted in the Inpatient Psychiatry Service. Patients will receive up to 6 ketamine or placebo infusions until, for 3 consecutive sessions, they have a clinician rated Scale for Suicidal Ideation (SSI) score of<4, and >50% decrease from baseline, and clinical assessment of patient not being suicidal, or they have been discharged from the inpatient unit. Patients will participate in weekly sessions of Collaborative Assessment for the management of Suicidality (CAMS), from the first week of the study while admitted to the hospital and will continue it on a weekly basis post-discharge until the patient has three consecutive outpatient CAMS sessions with an overall risk < 2 (# 6 on the SSF Core Assessment) along with a positive response regarding their thoughts/feelings and clinician indicating behavioral stability (suicidal behavior).

DETAILED DESCRIPTION:
Suicide is the second leading cause of death in 15-24 year-olds and accounts for 13% of all adolescent deaths annually. According to the CDC, the suicide rate for 10-24 year-olds increased in the last decade, with the suicide rate for 10-14 year-olds, 15-18 year-olds, and 20-24 year-olds increasing 177%, 76%, and 36%, respectfully. There is a critical need to develop fast and effective treatment in this highest-risk age group. Therefore, there is an urgent need to develop rapid, safe and feasible treatment to decrease suicidality in youth admitted to inpatient psychiatry after a serious suicidal attempt.

This proposal seeks to address this critical clinical gap by conducting an inpatient trial of treatment with ketamine vs placebo (saline) for rapid reversal of patients' suicidal state. Furthermore, this study will also test whether ketamine facilitates the effectiveness of collaborative psychotherapy for an enduring anti-suicidal response. One hundred and forty subjects who are medically stable admitted to inpatient psychiatry after a serious suicide attempt (defined as any act of self-harm with an intent to die) with continued suicidal ideation will be included in the study. After initial assessment, in conjunction with an anesthesiologist for any contraindication of using ketamine, patients will be randomized to receive either ketamine infusion 0.5 mg/kg over 40 minutes or saline. Ketamine or saline infusions on alternate days over two weeks will be given until subject reports no suicidal ideation for three consecutive sessions, or a maximum administration of six infusions is reached, or until they are discharged from the hospital. Concurrently, weekly sessions of CAMS will be started and continued as an outpatient after the patient is discharged until the subject also reports no suicidal ideation as an outpatient for three consecutive sessions. Monthly assessments for suicidal ideation, attempts and readmissions will be conducted as an outpatient for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 14 to 30 years of age
* Subjects must have been admitted to Cleveland Clinic Hospital (Fairview, Marymount, or Lutheran Hospital) or Massachusetts General Hospital (Blake 11) after a suicide attempt (any intentional, non-fatal self- injury regardless of medical lethality, if intent to die was indicated) with continued suicidal ideation or endorsing ongoing suicidal ideation and unable to contract for safety placing them at an increased risk to attempt suicide. Subjects will need a clinical rated Scale for Suicidal Ideation (SSI) score ≥ 6.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects with known history of autistic spectrum disorder; non-verbal patients.
* Subjects with moderate or severe intellectual disability (IQ less than 70 and those patients in special education full-time).
* Subjects with schizophrenia or history of any type of psychosis including mood disorder related psychosis and brief reactive psychosis.
* Within 6 months before initial screening, urine toxicology positive for phencyclidine, cocaine or amphetamines (subjects prescribed amphetamines for management of ADHD will not be excluded)
* Subjects with history of moderate or severe substance or alcohol use per DSM- V criteria in the past 6 months.
* Subjects with any contraindication to ketamine such as allergic reaction to ketamine or medical or neurological condition with a contraindication for use of ketamine or on any drugs associated with significant interaction with ketamine.
* Subjects who are currently pregnant and/or breast feeding.
* Subjects with previous recreational ketamine use. Subjects with previous therapeutic Ketamine use that exceeds the maximum cumulative lifetime exposure of 60 mg daily and 8 administrations maximum (or 480 mg) during both previous treatment and the proposed inclusion of this study.
* Subjects with hypertension, history of myocardial infarction, congestive heart failure of Stage 2 or higher, angina, or QTcF of at least 450 msec as indicated by chart review and/or standard of care EKG performed upon admission to inpatient unit.
* Subjects in the custody of Children's Services.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of remission of suicidal symptoms at the end of treatment. | Up to 3 months post-discharge
  Remission of suicide symptoms will be defined by a 50% or greater reduction in the clinician-rated baseline Beck Scale for Suicidal Ideation (SSI) score, and SSI score less than the score of 4. SSI scores can range from 0 to 38, and a higher score indicates increased severity of suicidal ideation. The primary outcome of the remission rate will be compared between the two groups.

SECONDARY OUTCOMES:
Number of CAMS sessions needed to achieve enduring mental state | Up to 3 months post-discharge
  Number of CAMS sessions needed to achieve enduring mental state
Change of Beck Scale for Suicide Ideation score will be analyzed | Up to 3 months post-discharge
  Change of Beck Scale for Suicide Ideation (SSI) score will be analyzed. SSI scores can range from 0 to 38, and a higher score indicates increased severity of suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Falcone, M.D., Principal Investigator — The Cleveland Clinic; Amit Anand, M.D., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Cleveland Clinic, Cleveland, Ohio